CLINICAL TRIAL: NCT00808912
Title: Decreased Pulmonary Artery Pressure by Oral Sildenafil Injection During Exercise in Air Pollution Increases Exercise Performance.
Brief Title: Does Sildenafil Increase Exercise Performance in Air Pollution?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marywood University (Other)
Responsible Party: Kenneth W. Rundell Ph.D., Marywood University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MU2007-028
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Pulmonary Hypertension; Pulmonary Artery Pressure; Exercise Performance; Air Pollution
Keywords: phosphodiesterase; sildenafil; pulmonary hypertension; exercise performance; air pollution
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Subjects will exercise in a high air pollutant environment after ingesting a standard dose of sildenafil.
  Interventions: Drug: sildenafil
- 2 (Active Comparator): Subjects will exercise in a low pollutant environment after ingesting a standard dose of sildenafil.
  Interventions: Drug: sildenafil
- 3 (Placebo Comparator): Subjects will exercise in a high pollutant environment after ingesting a placebo.
  Interventions: Other: placebo
- 4 (Placebo Comparator): Subjects will exercise in a low pollutant environment after ingesting a placebo.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: sildenafil — sildenafil 50 mg ingested orally 1 hour prior to exercise testing
  Other Names: Viagra
  Arms: 1; 2
Other: placebo — matching placebo for sildenafil 50 mg to be ingested orally 1 hour prior to exercise testing.
  Other Names: sugar pill
  Arms: 3; 4

SUMMARY:
The purpose of this study is to examine if the ingestion of a standard dose of sildenafil enhances the athletic performance of competitive athletes when exercising in a high pollutant environment verses a low air pollutant environment.

DETAILED DESCRIPTION:
This study will evaluate effects of sildenafil on exercise performance while breathing high levels of emission exhaust ultrafine and fine particulate matter. Exercise performance will be measured by work accumulation (total kJ) during a 6-min maximal effort cycle ergometer ride (CER) done immediately after 30 min cycling at 75% of 6 min mean watts determined from familiarization trial. Peak oxygen consumption, cardiac output, pulmonary artery pressure, diffusion capacity(DLco), and SaO2 will be determined for each trial. Blood and urine will be analyzed for sildenafil using LC/MS.

ELIGIBILITY:
Inclusion Criteria:

* non-asthmatic
* asthmatic
* active participants in endurance sports.

Exclusion Criteria:

* history of high blood pressure
* history of heart disease
* pulmonary arterial hypertension
* pulmonary emboli
* diagnosis of moderate to severe asthma (FEV1 <75% predicted)
* pregnant or lactating

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
That a decrease in exercise performance subsequent to emissions particle inhalation will be blunted by oral ingestion of 50 mg sildenafil prior to a 6-min maximal accumulation test (total kJ)on a cycle ergometer. | Cycle ergometer testing will be done one hour after administration of sildenafil or matching placebo.

SECONDARY OUTCOMES:
That the decreased VO2 peak and decreased exercise performance from emissions inhalation will be the result of pulmonary hypertension causing decreased stroke volume. | Pulmonary artery pressure will be measured before and immediately post exercise.
That plasma and urine sildenafil and metabolites will be measurable by liquid chromatography mass spectrometry (LC/MS) 6 h post ingestion. | Blood and urine samples will be collected at 1, 3, 1nd 6 hours post exercise testing.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Rundell, Ph.D., Principal Investigator — Marywood University
Locations (1):
- Marywood University, Scranton, Pennsylvania, United States